CLINICAL TRIAL: NCT02120027
Title: A 52-Week, Double-blind, Randomised, Placebo-controlled, Parallel-group Phase III Study With Re-randomisations at Week 25 to Evaluate the Efficacy and Safety of Oral Ibodutant 10 mg Once Daily in Female Patients With Irritable Bowel Syndrome With Diarrhoea (IBS-D)
Brief Title: 52-Week Efficacy and Safety Study of Ibodutant in Women With Irritable Bowel Syndrome With Diarrhea (IBS-D)
Acronym: IRIS-4
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Because of negative results of the sister study NAK-06 and the low overall response rate at week 24.
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAK-07; 2013-000895-14 (EudraCT Number)
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: Irritable Bowel Syndrome; Colon, irritable; Bowel disease; Diarrhea
MeSH Terms: conditions — Irritable Bowel Syndrome; Intestinal Diseases; Diarrhea | interventions — ibodutant; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibodutant 10 mg (Experimental): Oral tablet to be given once daily for 24 weeks of treatment. Patients randomised to the ibodutant 10 mg arm will continue on ibodutant 10 mg for additional 28 weeks of treatment via mock-re-randomisation at week 25 .
  Interventions: Drug: Ibodutant 10 mg
- Placebo (Placebo Comparator): Oral tablet to be given once daily for 24 weeks of treatment. Patients randomised to the placebo arm will be re-randomised at week 25 in a 1:1 ratio to ibodutant or placebo for additional 28 weeks of treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibodutant 10 mg — Oral tablet, to be given once daily.
  Other Names: Code: MEN 15596
  Arms: Ibodutant 10 mg
Drug: Placebo — Oral tablet (identical in appearance and weight to ibodutant tablets) to be given once daily.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Irritable Bowel Syndrome with diarrhoea (IBS-D) is a functional gastrointestinal disorder characterised by chronic or recurrent abdominal pain or discomfort and diarrhoea. This trial aims at the evaluation of the efficacy and safety of oral ibodutant 10 mg once daily as compared to placebo in women with IBS-D over a 24-week treatment period.

DETAILED DESCRIPTION:
The study evaluates the efficacy and safety of ibodutant 10 mg, given once daily for 24 weeks in comparison with placebo in female IBS-D patients. Randomisation to ibodutant and placebo will be 1:1. Efficacy is evaluated in terms of weekly response for abdominal pain intensity and stool consistency over 24 weeks of treatment in at least 50% of the weeks of treatment.

The clinical phase of the study comprises up to 2 weeks of screening for patient's eligibility, a 2-week run-in period (treatment-free) for IBS severity assessment, a first 24-week double-blind treatment period, a second 28-week re-randomised double-blind treatment period and a 2-week safety follow-up, resulting in a maximum 58-week overall duration of the study for each patient.

Patients report their IBS-related symptoms daily in a telephone-based electronic diary from run-in until end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* At screening:

  * Female patients aged 18 years or older.
  * Clinical diagnosis of IBS-D according to the following symptoms-based criteria as per Rome III modular questionnaire criteria:

    1. Recurrent abdominal pain or discomfort for at least 3 days per month in the last 3 months associated with at least 2 of the following characteristics: a) improvement with defecation; b) onset associated with a change in the frequency of stool; c) onset associated with a change in form (appearance) of stool.
    2. Symptom-onset at least 6 months prior to diagnosis.
    3. Loose or watery stools at least 25% of the time in the last 3 months AND hard or lumpy stools less than 25% of the time in the last 3 months.
    4. Additional criterion: more than 3 bowel movements per day at least 25% of the time in the last 3 months.
  * For patients older than 50 years OR patients with a positive family history of colorectal cancer: normal results from colonoscopy/flexible sigmoidoscopy performed within the last 5 years.
  * For patients aged 65 years or older: absence of ischaemic colitis, microscopy colitis or any other organic gastrointestinal disease as evidenced by the results of a colonoscopy/flexible sigmoidoscopy with biopsy performed within 6 months.
  * For women of childbearing potential: Use of a highly effective contraceptive method with a failure rate <1% per year throughout the entire study period.
  * Physical examination without clinically relevant abnormalities during screening.
  * No clinically relevant abnormalities in 12-Lead ECG or in laboratory findings.
  * Mentally competent, able to give written informed consent, and compliant to undergo all visits and procedures.
  * Unrestricted access to a touch-tone telephone.
  * Willingness to refrain from using loperamide within 3 days prior to run-in visit and during the run-in period.

Additional criteria at randomisation:

* During both weeks of the run-in period:

  1. A weekly average of worst abdominal pain in the past 24 hours with a score of ≥3.0 on a 0 to 10 point scale.
  2. At least one bowel movement on each day.
  3. A weekly average of at least 3 bowel movements per day.
  4. At least one stool with a consistency of Type 6 or Type 7 according to the Bristol Stool Scale (BSS) on at least 2 days per week.
  5. Less than 2 bowel movements with a consistency of Type 1 or Type 2 according to the BSS per week.
  6. Adequate compliance with the e-diary recording procedure defined as at least 11 of 14 days (≥75%) of the nominal daily data entry.

     Exclusion Criteria:
* Male gender.
* Diagnosis of IBS with a subtype of constipation, mixed IBS, or un-subtyped IBS.
* Colonic or major abdominal surgery, any other major abdominal surgery or elective major surgery planned or expected during the study.
* History of organic GI abnormalities, inflammatory bowel diseases, complicated diverticulosis, ischaemic colitis, microscopic colitis.
* History of pancreatitis, active biliary duct disease, cholecystitis or symptomatic gallbladder stone disease in the previous 6 months.
* History of gluten enteropathy or lactose intolerance.
* Current or previous diagnosis of neoplasia.
* History of endometriosis.
* History of positive tests for ova or parasites, or clostridium difficile toxin or occult blood in the stool in the previous 6 months.
* History of human immunodeficiency virus infection.
* History of major cardiovascular events in the previous 6 months.
* Uncontrolled hypertension, insulin-dependent diabetes mellitus or abnormal thyroid function.
* Major psychiatric or neurological disorders or unstable medical condition which may compromise the efficacy and safety assessments.
* Evidence of clinically significant hepatic disease, severe renal insufficiency or anemia.
* Relevant changes in dietary habits, lifestyle, or exercise regimen in the previous 2 months.
* Use of prohibited concurrent medication within the previous month such as antibiotics, antimuscarinic drugs, drugs enhancing GI motility and analgesics.
* Pregnancy or breastfeeding.
* Inability to understand or collaborate throughout the study.
* Participation in other clinical studies in the previous 4 weeks or concurrent enrollment in a clinical study.
* Any condition that would compromise the well-being of the patient.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Professor, Study Chair — Department of Gastroenterology, University Hospital Gasthuisberg, Katholieke Universiteit Leuven, Leuven, Belgium; Lin Chang, Professor, Study Chair — Digestive Health and Nutrition Clinic. University of California, Los Angeles, CA, USA
Locations (119):
- United States (65):
  - Chandler, Arizona
  - Glendale, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - North Little Rock, Arkansas
  - Encino, California
  - Gold River, California
  - Laguna Hills, California
  - Lincoln, California
  - North Hollywood, California
  - Orange, California
  - Pasadena, California
  - San Diego, California
  - Centennial, Colorado
  - Colorado Springs, Colorado
  - Fort Myers, Florida
  - Hialeah, Florida
  - Inverness, Florida
  - Kissimmee, Florida
  - Lauderdale Lakes, Florida
  - Miami, Florida
  - Miami Lakes, Florida
  - Pinellas Park, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - Addison, Illinois
  - Oak Lawn, Illinois
  - Rockford, Illinois
  - Evansville, Indiana
  - Clive, Iowa
  - Shawnee, Kansas
  - Metairie, Louisiana
  - Shreveport, Louisiana
  - Columbia, Maryland
  - Brockton, Massachusetts
  - Wyoming, Michigan
  - St Louis, Missouri
  - Billings, Montana
  - Newington, New Hampshire
  - Brooklyn, New York
  - Great Neck, New York
  - New York, New York
  - Hickory, North Carolina
  - High Point, North Carolina
  - Kinston, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Franklin, Ohio
  - Mentor, Ohio
  - Levittown, Pennsylvania
  - Anderson, South Carolina
  - Germantown, Tennessee
  - Jackson, Tennessee
  - Kingsport, Tennessee
  - Arlington, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Logan, Utah
  - Ogden, Utah
  - Sandy City, Utah
  - Lynchburgh, Virginia
  - Seattle, Washington
  - Spokane, Washington
- Czechia (7):
  - České Budějovice
  - Hradec Králové
  - Kralove
  - Prague
  - Příbram
  - Slaný
  - Zlín
- Germany (9):
  - Berlin
  - Bochum
  - Frankfurt
  - Hamburg
  - Hanover
  - Karlsruhe
  - Leipzig
  - Mainz
  - Schwerin
- Hungary (7):
  - Budapest
  - Debrecen
  - Gyula
  - Mátészalka
  - Pécs
  - Szekszárd
  - Vác
- Latvia (4):
  - Daugavpils
  - Riga
  - Riga III
  - Valmiera
- Poland (7):
  - Katowice
  - Lodz
  - Poznan
  - Sopot
  - Staszów
  - Warsaw
  - Wroclaw
- Slovakia (5):
  - Bratislava
  - Ilava
  - Nitra
  - Trenčín
  - Trnava
- Sweden (4):
  - Gothenburg
  - Lund
  - Stockholm
  - Uppsala
- United Kingdom (11):
  - Bexhill-on-Sea
  - Chorley
  - Coventry
  - Edgbaston
  - Glasgow
  - Llanishen
  - North Manchester
  - Northumberland
  - Norwich
  - Reading
  - Waterloo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was screened on 26th February 2014 and the first patient randomised on 24th March 2014. The last patient completed the study on 03rd November 2015. The study was conducted at 139 clinical sites in 9 countries (Czech Rep, Germany, Hungary, Latvia, Poland, Slovakia, Sweden, the USA and the United Kingdom)
Pre-assignment Details: A total of 1300 patients entered a 2-week Screening period, 1072 entered the qualifying 2-week Run-in period and 558 of them were randomised. Two patients randomised to placebo never took the study medication.
Period: Overall Study
Arm/Group | Ibodutant 10 mg | Placebo
Started | 277 | 279
Completed | 161 | 160
Not Completed | 116 | 119
Not completed — Adverse Event | 4 | 5
Not completed — Lack of Efficacy | 3 | 5
Not completed — Lost to Follow-up | 5 | 13
Not completed — Other | 4 | 0
Not completed — Physician Decision | 4 | 3
Not completed — Protocol Violation | 18 | 21
Not completed — Study terminated by Sponsor | 45 | 47
Not completed — Withdrawal by Subject | 33 | 25

BASELINE CHARACTERISTICS:
Population: Baseline analysis was performed on the ITT population (n=556). The ITT population includes all randomised patients who took at least one dose of study drug.
Groups:
- Placebo: Oral tablet to be given once daily for 24 weeks of treatment. Patients randomised to the placebo arm will be re-randomised at week 25 in a 1:1 ratio to ibodutant or placebo for additional 28 weeks of treatment.
  Placebo: Oral tablet, (identical in appearance and weight to ibodutant tablets), to be given once daily.
- Total: Total of all reporting groups
Arm/Group | Ibodutant 10 mg | Placebo | Total
Number analyzed (Participants) | 277 | 279 | 556
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 269 | 269 | 538
  >=65 years | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (12.2) | 43.8 (11.8) | 43.2 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 277 | 279 | 556
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 124 | 131 | 255
  Not Hispanic or Latino | 153 | 148 | 301
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 28 | 60
  White | 241 | 247 | 488
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Geographic Region [Count of Participants; unit: Participants]
  Eastern Europe | 35 | 30 | 65
  North America | 211 | 214 | 425
  Western Europe | 31 | 35 | 66
Body Mass Index, Continuous [Mean (Standard Deviation); unit: kg/m²] | 29.6 (6.92) | 29.6 (7.02) | 29.6 (6.96)
Abdominal Pain Severity, Categorical [Count of Participants; unit: Participants] — Worst abdominal pain on a 0 to 10 scale, where 0 corresponds to no pain and 10 corresponds to worst possible pain.
  Participants
    Abdominal Pain Severity < 5 | 55 | 54 | 109
    Abdominal Pain Severity ≥ 5 and < 8 | 172 | 172 | 344
    Abdominal Pain Severity ≥ 8 | 50 | 53 | 103
IBS-Signs and Symptoms Score, Categorical [Count of Participants; unit: Participants] — IBS-SSS score calculated from the questionnaire evaluating primarily the intensity of IBS symptoms during a 10-day period in the following domains: abdominal pain, distension, bowel habits (stool frequency and consistency), and interference with life in general. The IBS-SSS calculates the sum of five items each scored on a visual analog scale from 0 to 100. All five items contribute equally to the total score, yielding a range of 0 to 500 to categorize patients into three severity groups: mild (below 175), moderate (175-300), and severe (above 300).
  Participants
    Mild IBS | 7 | 7 | 14
    Moderate IBS | 60 | 58 | 118
    Severe IBS | 210 | 214 | 424

OUTCOME MEASURES:

1. Primary Outcome: Weekly Response for Abdominal Pain Intensity AND Stool Consistency Over the First 24 Weeks of Treatment in at Least 50% of the Weeks of Treatment (12 Out of 24 Weeks).
Description: The patient will be considered a weekly responder if she meets both of the following criteria in the same week:
  * Abdominal pain response: decrease in weekly average of worst abdominal pain score in the past 24 hours of at least 30% compared with baseline (patients reported their worst abdominal pain on a 0 to 10 NRS scale, where 0 corresponds to no pain and 10 corresponds to worst possible pain);
  * Stool consistency response: decrease of at least 50% in the number of days per week with at least one stool that has a consistency of Type 6 or 7 compared with baseline (patients reported their stool consistency response using the Bristol Stool Chart score based on a 1 to 7 NRS scale where 1 corresponds to hard stool and 7 corresponds to watery diarrhoea).
Time Frame: 24 weeks
Population: Modified ITT (mITT) Population: all patients included in the ITT population excluding patients from site 00179 (N=48), where a potential serious breach of Good Clinical Practice was reported, and site 00186 (N=34), where disqualification proceedings against the Investigator were initiated by the US Food and Drug Administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibodutant 10 mg | Placebo
Number analyzed (Participants) | 236 | 238
Participants | 51 | 52
Statistical Analysis 1: Comparison: Ibodutant 10 mg vs Placebo; Test type: Superiority or Other; p = 0.949, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.986, 95% CI 2-sided [0.64 to 1.53]

2. Secondary Outcome: Weekly Response for Abdominal Pain Intensity Over the First 24 Weeks of Treatment in at Least 50% of the Weeks of Treatment (12 Out of 24 Weeks).
Description: The patient will be considered a weekly abdominal pain responder if she meets the following criterion:
  * Decrease in weekly average of worst abdominal pain score in the past 24 hours of at least 30% compared with baseline.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ibodutant 10 mg | Placebo
Number analyzed (Participants) | 236 | 238
Participants | 96 | 83
Statistical Analysis 1: Comparison: Ibodutant 10 mg vs Placebo; Test type: Superiority or Other; p = 0.193, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.280, 95% CI 2-sided [0.88 to 1.86]

3. Secondary Outcome: Weekly Response for Stool Consistency Over the First 24 Weeks of Treatment in at Least 50% of the Weeks of Treatment (12 Out of 24 Weeks).
Description: The patient was considered a weekly stool consistency responder if she met the following criterion:
  * Decrease of at least 50% in the number of days per week with at least one stool that has a consistency of Type 6 or 7 compared with baseline.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ibodutant 10 mg | Placebo
Number analyzed (Participants) | 236 | 238
Participants | 72 | 71
Statistical Analysis 1: Comparison: Ibodutant 10 mg vs Placebo; Test type: Superiority or Other; p = 0.872, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.032, 95% CI 2-sided [0.70 to 1.53]

4. Secondary Outcome: Weekly Response for Relief of Overall IBS Signs and Symptoms Over the First 24 Weeks of Treatment in at Least 50% of the Weeks (12 Out of 24)
Description: The patient was considered a weekly responder if she has an IBS degree-of-relief equal to "completely relieved/improved" or "considerably relieved/improved".
  Weekly e-diary assessment of IBS degree-of-relief of overall on signs or symptoms over the last 7 days was collected using a balanced 7-point Likert scale with 1= Completely relieved/improved, 2= Considerably relieved/improved, 3=Somewhat relieved/improved, 4= Unchanged, 5= Somewhat worse, 6=Considerably worse, 7= As bad as I can imagine.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ibodutant 10 mg | Placebo
Number analyzed (Participants) | 236 | 238
Participants | 37 | 29
Statistical Analysis 1: Comparison: Ibodutant 10 mg vs Placebo; Test type: Superiority or Other; p = 0.272, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.339, 95% CI 2-sided [0.79 to 2.26]

5. Secondary Outcome: Sustained Analysis of Response for Abdominal Pain AND Stool Consistency Over First 24-week Double-blind Treatment Period
Description: Weekly response for abdominal pain intensity AND stool consistency over the first 24 weeks of treatment in at least 50% of the weeks of treatment (12 out of 24 weeks) with at least 2 weeks of response in the last 4 weeks of treatment (week 21 to 24). The patient will be considered a weekly responder as defined for the primary endpoint.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ibodutant 10 mg | Placebo
Number analyzed (Participants) | 236 | 238
Participants | 50 | 45
Statistical Analysis 1: Comparison: Ibodutant 10 mg vs Placebo; Test type: Superiority or Other; p = 0.567, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.153, 95% CI 2-sided [0.73 to 1.81]

ADVERSE EVENTS:
Time Frame: Adverse Events were reported for the safety population (all enrolled patients who received at least 1 dose of study drug) over a period of 24 weeks (first 24-week double-blind treatment period).
Description: AEs were categorized as Treatment-Emergent Signs and Symptoms (TESS) or Non-TESS for each of the study periods based on the onset date/time of AE. Number of events and number of patients (%) are presented by System Organ Class (SOC) and Preferred Term (PT). All serious TESS are reported for patients in any arm for the first 24-week period. No change in incidence of serious TESS was observed over the entire 52-weeks of study treatment with respect to the first 24-week treatment period.
Groups:
- Ibodutant 10 mg for 24-week Treatment: Oral tablet to be given once daily for 24 weeks of treatment.
  Ibodutant 10 mg: Oral tablet, to be given once daily.
- Placebo for 24-week Treatment: Oral tablet to be given once daily for 24 weeks of treatment.
  Placebo: Oral tablet, (identical in appearance and weight to ibodutant tablets), to be given once daily.
Arm/Group | Ibodutant 10 mg for 24-week Treatment | Placebo for 24-week Treatment
Serious Adverse Events (participants affected / at risk) | 3/277 | 2/279
Other Adverse Events (participants affected / at risk) | 75/277 | 82/279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibodutant 10 mg for 24-week Treatment (N=277) | Placebo for 24-week Treatment (N=279)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Occipital neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoe (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibodutant 10 mg for 24-week Treatment (N=277) | Placebo for 24-week Treatment (N=279)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (4)
Nausea (Gastrointestinal disorders) | 7 (9) | 5 (5)
Gastroenteritis (Gastrointestinal disorders) | 6 (7) | 1 (1)
Nasopharyngitis (Infections and infestations) | 8 (9) | 19 (21)
Sinusitis (Infections and infestations) | 2 (2) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 4 (4)
Urinary tract infection (Infections and infestations) | 9 (9) | 9 (9)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (8) | 4 (4)
Headache (Nervous system disorders) | 3 (3) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 3 (3)
Fatigue (General disorders) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 3 (3)
Weight increased (Investigations) | 0 (0) | 3 (3)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Migraine (Nervous system disorders) | 4 (10) | 0 (0)

LIMITATIONS AND CAVEATS:
The Sponsor decided on 03 September 2015 to prematurely terminate the study because of negative results of the contemporaneous sister study NAK-06 and the definitely lower than expected overall (ibodutant/placebo) response rate at week 24.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting the results of this study for publication or presentation, the Investigator will allow the sponsor at least 30 days time to review and comment upon the publication manuscript. It is agreed, that the results of the study will not be submitted for presentation, abstract, poster exhibition, or publication by the investigator until Menarini Ricerche S.p.A. has reviewed/commented and agreed to any publication.